CLINICAL TRIAL: NCT06875505
Title: Post-activation Performance Enhancement in Soccer Players: The Effect of Different Contraction and Rest Periods on Changing Direction Ability
Brief Title: Post-activation Performance Enhancement in Soccer Players:
Acronym: PAPEsoccer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Neslihan AKÇAY, Assoc. Prof. Dr, Karabuk University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: UKarabuk-3
Record Dates: First submitted 2025-03-08; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Performance; Post Activation Potentiation; Soccer
Keywords: Soccer; Post activation Performance Enhancement; Dynamic Contraction; Isometric contraction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants were strictly separated and think their intervention is the main intervention. The same is true for care providers. Outcome assessors were unaware of participant group status and were not allowed to ask correspondingly.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dynamic PAPE (Experimental): In this protocol, the load determined for footballers during knee extension will be applied as 90% of their one repetition maximum (1TM). After the standard warm-up session at the beginning, the protocol will be performed by performing 1 set of 3 repetitions with the previously determined 1TM 90% load without resting between repetitions.
  Interventions: Other: Dynamic PAPE
- Isometric PAPE (Experimental): Isometric contraction will be used in the protocol. On the leg extension machine, the protocol will be performed by applying 3 sets of 3 seconds against only the lever arm with 1TM 90% load, 2 minutes rest will be applied between sets.
  Interventions: Other: Isometric PAPE

INTERVENTIONS:
Other: Dynamic PAPE — In this protocol, the load determined for footballers during knee extension will be applied as 90% of their one repetition maximum (1TM). After a standard warm-up session at the beginning, the protocol will be performed by performing 1 set of 3 repetitions with the previously determined 1TM 90% load without resting between repetitions. Isometric knee extension exercise will be used in the protocol. The movement will be performed sitting, in a position suitable for limb lengths and in a controlled manner using a leg extension machine. At the beginning of the movement, the knees will be flexed 90° and the adjustable lever arm of the machine will be fixed at this angle. Then they will be asked to perform bilateral isometric knee extension until the knees form a 180° angle. They will also be verbally motivated to complete the knee extension exercise.
  Arms: Dynamic PAPE
Other: Isometric PAPE — Isometric contraction will be used in the protocol. On the leg extension machine, the protocol will be performed by applying 3 sets of 3 seconds against the lever arm only with 1TM 90% load, 2 minutes rest will be applied between sets. Isometric knee extension exercise will be used in the protocol. The movement will be performed sitting, in a position suitable for limb lengths and in a controlled manner using a leg extension machine. At the beginning of the movement, the knees will be flexed 90° and the adjustable lever arm of the machine will be fixed at this angle. Then they will be asked to perform bilateral isometric knee extension until the knees form a 180° angle. They will also be verbally motivated to complete the knee extension exercise.
  Arms: Isometric PAPE

SUMMARY:
This study will be conducted in a randomised, crossover design. Soccer players will participate in two test sessions 48 hours apart. The athletes will be pre-tested in the professional direction change test and after the PAPE protocol of the group they are included in is applied, they will be taken to the professional direction change test at 15th second, 3rd, 6th, 9th and 12th minutes.

DETAILED DESCRIPTION:
This study will be conducted in a randomised, crossover design. Subjects will participate in two test sessions 48 hours apart. To eliminate the effect of fatigue, participants will be warned not to engage in intense physical activity before the study days and to pay attention to adequate carbohydrate intake so that repeated sprint performance will not be affected. On the 1st day of the study, after the participants were informed about the study, their heights will be recorded with a height meter, and their weights and body fat percentages will be taken with the Inbody 270 device. After the descriptive characteristics of all participants are obtained, the warm-up protocol will be applied and 1 RM will be determined and recorded by performing knee extension movement on the Knee Extension device. On the second day of the study, all athletes will be pre-tested in the professional change of direction test and will be taken to the professional change of direction test at 15 seconds, 3 minutes, 6 minutes, 9 minutes and 12 minutes after the PAPE protocol of the group they are included in is applied. On the third day of the study, the pre-tests of all athletes in the professional direction change test will be taken again and they will be taken to the professional direction change test at 15 seconds, 3rd, 6th, 9th and 12th minutes after the PAPE protocol of the group they are included in is applied. Participants will be asked to stop eating 1.5 hours before the measurement time. Athletes will be allowed to drink water (500ml) during the test and will be verbally motivated during the professional change of direction test.

ELIGIBILITY:
Inclusion Criteria:

* Being healthy
* Male soccer players
* Willing to maintain the intervention for all sessions

Exclusion Criteria:

* Under 18 years of age
* Having a chronic disease
* Contraindications for exercise

Ages: 18 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-04-25 (Estimated)

PRIMARY OUTCOMES:
Significant difference in dynamic condition | From baseline to the end of measurement at 1 weeks
  It is expected that there will be a significant difference in the rate of change of direction during different rest periods in the dynamic contraction condition compared to the isometric contraction condition
Significant difference in isometric condition | From baseline to the end of measurement at 1 weeks
  It is expected that there would be a significant difference in the rate of direction change during different rest periods in the isometric contraction condition compared to the dynamic contraction condition.
The time between the conditions is different | From baseline to the end of measurement at 1 weeks.
  Compared to the first measurement, a change in the rate of directional change in conditions is expected.

OTHER OUTCOMES:
Anthropometric Measurements 1 | Baseline
  Participants' height (cm) will assess by using a stadiometer (Holtain Stadiometer, England)
Anthropometric Measurements 2 | Baseline
  Body weight (kg) will asses by Inbody 270 (Biospace, California, USA).
Anthropometric Measurements 3 | Baseline
  Body mass index (BMI) (kg/m2) will asses by Inbody 270 (Biospace, California, USA).
Anthropometric Measurements 4 | Baseline
  Body fat percentage (%) will asses by Inbody 270 (Biospace, California, USA).
Knee Extension 1Repetition maximum Test | Baseline
  The 1RM of the soccer players will be performed on the leg extension device. The warm-up will be followed by a standard warm-up set of five repetitions with 50% of their estimated 1RM. Following this, participants will complete a preparation phase of 1-2 sets of 2-3 repetitions with a load corresponding to approximately 60-80% of their estimated 1RM.

CONTACTS AND LOCATIONS:
Overall Officials: Neslihan Akçay, Study Chair — Karabuk University
Locations (1):
- Karabuk University, Karabük, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Marshall J, Turner AN, Jarvis PT, Maloney SJ, Cree JA, Bishop CJ. Postactivation Potentiation and Change of Direction Speed in Elite Academy Rugby Players. J Strength Cond Res. 2019 Jun;33(6):1551-1556. doi: 10.1519/JSC.0000000000001834. PMID 28166184
- [Background] Keskin K, Akcay N, Ozmen T, Contarli N, Yildiz KC, Sofuoglu C, Kamis O, Rolnick N, de Queiros VS, Montoye A. Effects of different pre-exercise strategies on jumping performance in female volleyball players. J Sports Med Phys Fitness. 2025 Jan;65(1):59-68. doi: 10.23736/S0022-4707.24.16196-8. Epub 2024 Oct 3. PMID 39360986